CLINICAL TRIAL: NCT03688919
Title: Targeting Self-regulation to Promote Adherence and Health Behaviors in Children
Brief Title: Adolescent Interventions to Manage Self-regulation of T1D (AIMS T1D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Miller, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UH3HD087979 (NIH); UH3HD087979 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-28 (Actual); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Self-regulation; Medication Adherence
Keywords: adolescents; Type 1 Diabetes
MeSH Terms: conditions — Self-Control; Medication Adherence; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison (No Intervention): Adolescents and their families in this group will not receive any of the interventions.
- Self-Regulation Intervention (Experimental): This arm will use a computer-based working memory training game (NBack) targeting Executive Functioning and in-person relaxation and biofeedback training targeting Emotion Regulation. As well, adolescents will receive Future Orientation training by being asked to envision and describe future events they are looking forward to, using concrete, vivid descriptive language.
  Interventions: Behavioral: Self-Regulation Intervention

INTERVENTIONS:
Behavioral: Self-Regulation Intervention — The intervention targets Executive Functioning (EF), Emotion Regulation (ER) and Future Orientation (FO). The intervention will occur through home practice and text based reminders and mobile apps to practice techniques. For EF, youth will use the NBack intervention, a computer-based working memory training game. For ER, participants will engage in relaxation and biofeedback activities by completing activities (e.g., modulating breathing to keep heart rate) while wearing sensors. For FO, participants will envision and describe future events they are looking forward to, using concrete, vivid descriptive language. These descriptions will be audio recorded so that the participant can play back the cues at home at specified times of day (e.g., 7am and 3:30PM).
  Arms: Self-Regulation Intervention

SUMMARY:
This goal of this project is to test whether self-regulation assays and interventions can be delivered and change self-regulation in a sample of adolescents, specifically to test in a small randomized clinical trial (RCT) whether self-regulation interventions lead to change in medication adherence. The study will focus on adolescents with Type 1 Diabetes (T1D). These youth have clear medication adherence goals, yet are often non adherent and at great health risk during this developmental period. As responsibility for diabetes management shifts from parent to youth during this time, intervening with adolescents directly is vital for prevention.

DETAILED DESCRIPTION:
The goal of this study is to test whether interventions change self-regulation (SR) targets most relevant for medication adherence in youth with Type 1 Diabetes (T1D). Poor self-regulation has been identified in youth with T1D and is proposed as a central mechanism contributing to high rates of nonadherence and thus long-term complications, in pediatric T1D populations, particularly adolescents. As responsibility for T1D management shifts from parent to youth during this time, addressing self-regulation in adolescence is critical.

The study's self-regulation targets are executive functioning (EF; working memory, inhibitory control); emotion regulation (ER; capacity to manage stress, worry), and future orientation (FO; capacity to focus on future goals). The investigators posit that these self-regulation capacities are critical in order to engage in the multiple adherence behaviors (e.g., self-monitoring blood glucose, administering insulin via daily injections or a pump, regulating carbohydrate intake, physical activity, minimizing hyper-/hypo-glycemia) youth must follow to achieve and maintain optimal glycemic control. Thus, in addition to targeting T1D-specific adherence, it is essential to employ an experimental medicine approach to test whether improving self-regulation results in improved adherence behaviors and T1D-related health outcomes (quality of life; HbA1C). Yet, these self-regulation targets have not been rigorously tested as mechanisms of behavior change to improve adherence to T1D regimens in youth.

Using previously developed multimethod assays of these targets, the investigators will test the impact of interventions on these self-regulation targets, medical regimen adherence behaviors, and diabetes-related health outcomes (quality of life; HbA1C) in youth. The Scientific Premise is that poor self-regulation underlies poor medical regimen adherence. If improving self-regulation targets increase adherence in youth with T1D this approach may apply to other youth who must manage medical regimens. Findings will thus not only inform understanding of self-regulation as a mechanism of behavior change but will generate novel intervention strategies that may have trans-diagnostic implications and broad impact. As interventions to be delivered are designed to be light-touch and scalable, they may yield useful tools to use in future studies of behavior change mechanisms. The investigators propose an RCT design to test the following Specific Aims in a sample of youth with T1D (ages 13-17 years, n=94):

Aim 1. Test the hypothesis that the interventions developed in a prior study (NCT03060863) enhance identified self-regulation targets (EF, ER, FO) in a population of adolescents with T1D.

Aim 2. Test whether interventions improve medical regimen adherence behaviors and T1D health outcomes.

Exploratory Aim. Examine whether parents' SR modifies the effects of the UH3's bundled intervention to improve youth SR on youth treatment regimen adherence.

ELIGIBILITY:
Inclusion Criteria:

* youth must have been diagnosed with T1D for at least 6 months;
* reside with a parent;
* have HbA1c>=7.0;
* regular access to WiFi; and
* feel comfortable speaking English enough to complete study activities; and

Exclusion Criteria:

* non-fluency in English in parent or youth;
* psychiatric or cognitive conditions (e.g., clinically significant depression assessed via phone screen at intake) that would impede ability to participate.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Miller, Ph.D., Principal Investigator — University of Michigan; Emily Fredericks, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication would be made available upon reasonable request.
Time Frame: IPD that underlie results in a publication would be made available 6 months after publication upon reasonable request.
Access Criteria: The PIs will review all requests for IPD.

REFERENCES:
- [Derived] Choe A, Fredericks EM, Albright D, Lee JM, Sturza JM, Riley HO, Kaciroti N, Bauer KW, Miller AL. Executive Functioning, Diabetes Distress, and Diabetes Management Among Adolescents With Type 1 Diabetes: Youth and Parent Perspectives. Pediatr Diabetes. 2025 Feb 27;2025:7036544. doi: 10.1155/pedi/7036544. eCollection 2025. PMID 40303942
- [Derived] Miller AL, Lo SL, Albright D, Lee JM, Hunter CM, Bauer KW, King R, Clark KM, Chaudhry K, Kaciroti N, Katz B, Fredericks EM. Adolescent Interventions to Manage Self-Regulation in Type 1 Diabetes (AIMS-T1D): randomized control trial study protocol. BMC Pediatr. 2020 Mar 7;20(1):112. doi: 10.1186/s12887-020-2012-7. PMID 32145739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youth with Type 1 Diabetes were recruited from pediatric endocrinology clinics in Michigan.
Period: Overall Study
Arm/Group | Comparison | Self-Regulation Intervention
Started | 41 | 47
Completed | 38 | 46
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — withdrawn by study team due to poor data validity | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparison | Self-Regulation Intervention | Total
Number analyzed (Participants) | 41 | 47 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 47 | 88
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.3) | 15.4 (1.5) | 15.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 21 | 26 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 38 | 46 | 84
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 36 | 39 | 75
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 47 | 88
Youth Executive Function (behavioral) [Mean (Standard Deviation); unit: z-score] — Behavioral EF is measured using standard tasks (Forward/Backward Digit Span, Go No Go; see outcome measures for additional description). A composite variable indicating better EF (i.e. correct Digit Span responses, faster/more accurate Go No Go responses) is generated by creating standardized z-scores for each task variable and calculating a mean score. The final variable analyzed will be the composite z-score that represents behavioral EF, scored such that higher scores indicate better EF and with a Z-score of 0 representing the population mean. Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  z-score
    number analyzed (Participants) | 38 | 46 | 84
    (all) | 0.00 (0.09) | 0.01 (0.08) | 0.00 (0.07)
Youth Executive Function (parent/child report) [Mean (Standard Deviation); unit: z-score] — Youth EF-report is assessed using parent- and self-reports on Behavior Rating Inventory of Executive Functioning, 2nd Ed. (BRIEF-2), a standardized measure assessing EF difficulties (e.g., trouble controlling impulses, paying attention). Three indices are calculated (Behavioral, Emotional, Cognitive Regulation) and combined to form a standardized Global Executive Composite (GEC; range 0-100). The final variable analyzed is a composite z-score averaging youth- and parent-reported GEC scores, scored such that higher scores indicate poorer EF and a Z-score of 0 representing the population mean. Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  z-score
    number analyzed (Participants) | 40 | 47 | 87
    (all) | -0.01 (0.12) | 0.03 (0.11) | 0.01 (0.08)
Youth Emotion Regulation (parent/child report) [Mean (Standard Deviation); unit: z-score] — ER will be measured based on parent- and youth self-reports on NIH Toolbox Perceived Stress Survey (PSS); youth-reported dysregulated affect based on Structured Interview for Disorders of Extreme Stress (SIDES); and youth-reported emotion experiences on Positive and Negative Affect Schedule (PANAS; see Outcome Measures for more detail). The final variable analyzed will be a composite z-score created by standardizing and averaging parent and youth reports on the PSS, SIDES, and PANAS, scored such that higher scores indicate worse ER and with a Z-score of 0 representing the population mean.
  z-score | 0.08 (0.12) | 0.02 (0.08) | 0.05 (0.07)
Youth Self Efficacy (parent/child report) [Mean (Standard Deviation); unit: z-score] — Youth self-efficacy is an aspect of Future Orientation (FO) that will be measured using a composite of the NIH Toolbox Self-Efficacy parent and youth report scales. Participants respond to questions about their child's or their own (in the case of the child) self-efficacy. Higher scores are indicative of greater perceived self-efficacy. The final variable analyzed will be a composite z-score representing youth self-efficacy, a standardized average of youth and parent reports scored such that higher scores indicate better Self-efficacy and with a Z-score of 0 representing the population mean.
  z-score | -0.21 (0.12) | 0.02 (0.11) | -0.09 (0.08)
Youth Future Orientation (child self report) [Mean (Standard Deviation); unit: z-score] — Considering the future and how one's actions can affect future consequences is an aspect of youth Future Orientation (FO) measured using Consideration of Future Consequences Scale. Higher scores indicate a greater consideration of future consequences or forward looking behavior. The final variable analyzed will be a z-score that represents self-reported FO, scored such that higher scores indicate better FO and with a Z-score of 0 representing the population mean. Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  z-score
    number analyzed (Participants) | 40 | 46 | 86
    (all) | -0.06 (0.17) | -0.15 (0.15) | -0.11 (0.11)
Youth Future Orientation (behavioral) [Mean (Standard Deviation); unit: z-score] — Discounting the future is an aspect of youth Future Orientation (FO) that will be objectively measured using 5-trial Delay Discounting Task (see Outcome measures for more details). Participants are asked whether they would prefer to receive an amount of money later or in or half the amount now; this process is repeated varying length of delay to generate a delay discounting curve. The final variable analyzed will be a z-score that represents the steepness of the discounting curve (rate); higher scores indicate poorer FO and a Z-score of 0 represents the population mean. Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  z-score
    number analyzed (Participants) | 37 | 44 | 81
    (all) | -0.12 (0.11) | -0.14 (0.19) | -0.13 (0.41)
Blood Glucose Monitoring [Count of Participants; unit: Participants] — Change in blood glucose monitoring (BGM) frequency assessed by downloading data from the prior two weeks from the adolescent's glucometer. Adherence to BGM is defined as an average of 4 blood glucose measurements/day. Note, changes in clinical care resulted in only 30% of the sample with BGM data; 70% of the sample had Continuous Glucose Monitors [CGM]). Thus, we used the data from self-reported monitoring or CGM use, measured by youth self-report on a Type 1 Diabetes adherence measure administered to all patients in the clinic that has been linked to HbA1c level (Lee et al., 2021). Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  Participants
    number analyzed (Participants) | 40 | 47 | 87
    (all) | 40 | 43 | 83
Insulin Administration Adherence [Count of Participants; unit: Participants] — Insulin administration adherence is defined as at least 3 short acting insulin boluses/day vs not. This is measured by youth self-report on a Type 1 Diabetes adherence measure administered to all Type 1 Diabetes patients in the clinic and has been linked to Hemoglobin A1c (HbA1c), an indicator of blood glucose level (Lee et al., 2021). Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
  Participants
    number analyzed (Participants) | 36 | 37 | 73
    (all) | 35 | 34 | 69
Self Care Inventory-Revised (Adherence) [Mean (Standard Deviation); unit: z-score] — The Self-Care Inventory Revised (SCI-R) is a youth- and parent-report measure of multiple T1D self-care adherence behaviors (e.g., monitoring/recording glucose, administering/adjusting insulin, regulating meals/exercise, keeping appointments). The final variable analyzed will be the composite z-score that represents SCI-R adherence based on youth and parent reports (standardized and averaged), scored such that higher scores indicate better adherence and with a Z-score of 0 representing the population mean.
  z-score | -0.20 (0.13) | 0.05 (0.12) | -0.07 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Youth Executive Function (Behavioral EF) at 8 Weeks (Z-score)
Description: Behavioral EF will be measured using standard tasks (Forward/Backward Digit Span, Go No Go). In Digit Span, subjects repeat numbers presented aloud in order or reverse order (8 questions of 2 trials each; correct response is 1 point; incorrect or no response is 0 points). Scores are summed for each trial; maximum total raw score is 16 points. In Go No Go, subjects hit a key to respond when they see the 'go' stimulus (presented for 300 ms) but not when they see the no-go stimulus. Go No Go responses are scored based on reaction time (seconds) and accuracy (0-100%). Then, we will generate a composite variable indicating better EF (i.e. correct Digit Span responses, faster/more accurate Go No Go responses) by creating standardized z-scores for each task variable and calculating a mean score. The final variable analyzed will be the composite z-score that represents behavioral EF, scored such that higher scores indicate better EF and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 30 | 38
z-score | 0.02 (0.07) | -0.02 (0.06)

2. Primary Outcome: Change From Baseline in Youth Executive Function (EF-report by Parent and Self) at 8 Weeks (Z-score)
Description: Youth EF-report will be assessed using parent- and self-report versions of The Behavior Rating Inventory of Executive Functioning, 2nd Edition (BRIEF-2), a standardized EF measure. Items assess ability to control impulses, pay attention, modulate responses, and anticipate events. Three broad indices are calculated (Behavior Regulation, or ability to control behavioral impulses; Emotion Regulation, or ability to control emotional reactions; and Cognitive Regulation, or ability to focus, pay attention, stay organized) and combined to form a Global Executive Composite (GEC) score, which is a standardized score representing overall EF difficulty (range 0-100). Youth and parent GEC scores are averaged to represent overall Global Executive Functioning. The final variable analyzed will be the composite z-score that combines youth- and parent-reported EF, scored such that higher scores indicate poorer EF and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
z-score | 0.04 (0.06) | -0.08 (0.05)

3. Primary Outcome: Change From Baseline in Youth Emotion Regulation (ER-report by Parent and Self) at 8 Weeks (Z-score)
Description: ER will be measured using a composite measure of parent- and self-reports on the NIH Toolbox Perceived Stress Survey, a 10-item measure of stress in children (items are summed to indicate greater perceived stress; range: 0-40); youth self-reports of dysregulated affect using a 6-item scale based on the Structured Interview for Disorders of Extreme Stress (SIDES Affect Dysregulation Scale; items are averaged to indicate more affect dysregulation, range: 1-6); and youth reports of emotion experiences on the 20-item Positive and Negative Affect Schedule (PANAS; items are summed to indicate more negative [10 items] and fewer positive experiences [10 items]; range: 10-50). The composite ER measure will be created by standardizing and averaging PSS, SIDES, and PANAS scores. The final variable analyzed will be this composite z-score that represents ER, scored such that higher scores indicate worse ER and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
z-score | -0.10 (0.05) | 0.07 (0.05)

4. Primary Outcome: Change From Baseline in Youth Self-Efficacy (Parent- and Self-reported) at 8 Weeks (Z-score)
Description: Youth self-efficacy is hypothesized to promote future-oriented thinking, and is thus an aspect of Future Orientation that will be measured using a composite of the NIH Toolbox Self-Efficacy parent report form and the self-report form. Both forms consist of 10 items. Participants respond to questions about their child's or their own (in the case of the child) self-efficacy. Mean scores are generated; higher scores are indicative of greater perceived self-efficacy. The final variable analyzed will be the composite z-score that represents youth self-efficacy based on parent and youth report, standardized and averaged and scored such that higher scores indicate better Self-efficacy and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
z-score | 0.23 (0.09) | 0.06 (0.08)

5. Primary Outcome: Change From Baseline in Youth Future Orientation (Self-report) at 8 Weeks (Z-score)
Description: Considering the future and how one's actions can affect future consequences is an aspect of youth Future Orientation (FO) that will be measured using the Consideration of Future Consequences Scale. Youth will answer 14 questions (e.g., "I think about how things would be in days to come, and try to influence those things in my daily behavior") on a 7-point scale ranging from 1=Not at all like me to 7=Neutral. Higher scores indicate a greater consideration of future consequences or forward looking behavior. The final variable analyzed will be a z-score that represents self-reported FO, scored such that higher scores indicate better FO and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
z-score | 0.06 (0.17) | 0.11 (0.16)

6. Primary Outcome: Change From Baseline in Youth Future Orientation (Objective Measure) at 8 Weeks (Z-score)
Description: The degree to which one discounts the future is an aspect of youth Future Orientation (FO) that will be objectively measured using 5-trial Delay Discounting Task. Each 5-trial version of this task uses one monetary amount per trial (e.g., $1, 000; $1, 000, 000). Participants are asked on the first trial of the task whether they would prefer to receive that amount in three weeks or half that amount now. On the next trial the question is repeated but with a different time delay according to response on the previous trial. That is, a greater delay is presented on the next trial if the participant chose "now" on the previous trial, whereas a lesser delay is presented if the participant chose the later time on the previous trial. The dependent measure is the steepness of the delay discounting curve. The final variable analyzed will be the z-score that represents this discount rate; higher scores indicate poorer FO and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 28 | 38
z-score | 0.09 (0.12) | 0.03 (0.11)

7. Secondary Outcome: Change From Baseline in Number of Participants Conducting Blood Glucose Monitoring at 8 Weeks
Description: Change in blood glucose monitoring (BGM) frequency will be assessed by downloading data from the prior two weeks from the adolescent's glucometer. Adherence to BGM is defined as an average of 4 blood glucose measurements/day. Note, we had missing data for the downloads due to changes in clinical care since this measure was proposed (only 30% of the sample had only meters so were not recommended by their provider to download their meters in this way; 70% of the sample had Continuous Glucose Monitors (CGM). Thus, we used the data from self-reported monitoring or CGM use, measured by youth self-report on a Type 1 Diabetes adherence measure administered to all patients in the clinic that has been linked to HbA1c level (Lee et al., 2021).
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Count of Participants; unit: Participants
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
Participants | 38 | 42

8. Secondary Outcome: Change From Baseline in in Number of Participants With Insulin Administration Adherence at 8 Weeks
Description: Insulin administration adherence is defined as at least 3 short acting insulin boluses/day vs not. This is measured by youth self-report on a Type 1 Diabetes adherence measure administered to all Type 1 Diabetes patients in the clinic and has been linked to Hemoglobin A1c (HbA1c), an indicator of blood glucose level (Lee et al., 2021).
Time Frame: baseline and 8 weeks
Population: Some missing data from this measure could not be analyzed so the total number analyzed differs from the population
Measure: Count of Participants; unit: Participants
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 32 | 39
Participants | 31 | 36

9. Secondary Outcome: Change From Baseline in Self-Care Inventory Revised at 8 Weeks (Z-score)
Description: The Self-Care Inventory Revised (SCI-R) is a 14-item youth- and parent-report measure of multiple T1D self-care adherence behaviors. Items reflect main aspects of the T1D regimen, including: monitoring and recording glucose, administering and adjusting insulin, regulating meals and exercise, and keeping appointments. Respondents report on adherence behaviors on a 5-point scale (1="never do it"; 5="always do this as recommended without fail"; or N/A.). The final variable analyzed will be the composite z-score that represents SCI-R adherence based on youth and parent reports, standardized and averaged and scored such that higher scores indicate better adherence and with a Z-score of 0 representing the population mean.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Comparison | Self-Regulation Intervention
Number analyzed (Participants) | 38 | 46
z-score | 0.23 (0.09) | 0.12 (0.08)

ADVERSE EVENTS:
Time Frame: Study timeframe (8 weeks)
Description: regular reporting to the Institutional Review Board (IRB), based on participant report or medical record review
Arm/Group | Comparison | Self-Regulation Intervention
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/47
Serious Adverse Events (participants affected / at risk) | 3/41 | 1/47
Other Adverse Events (participants affected / at risk) | 3/41 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparison (N=41) | Self-Regulation Intervention (N=47)
Diabetic ketoacidosis (DKA) (Endocrine disorders) | 2 (2) | 1 (1) — Diabetic ketoacidosis (DKA), expected for condition of Type 1 Diabetes, not study related
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Hyperglycemia, expected for condition of Type 1 Diabetes, not study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparison (N=41) | Self-Regulation Intervention (N=47)
ER visit (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — ER visit for wrist pain, unrelated to study
cataract surgery (Eye disorders) | 0 (0) | 2 (2) — Cataract surgery (planned), unrelated to study
ER visit (General disorders) | 2 (2) | 1 (1) — ER visit, felt sick, unrelated to study

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic occurred in the middle of our study, and we did not enroll new participants or conduct in person visits from 3/13/20-8/24/20 due to University of Michigan policies. It is possible the intervention was impacted by the pandemic.

Youth also self-reported high adherence in their blood glucose monitoring and insulin administration at baseline, so this likely reduced our ability to find effects on these secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT03688919/Prot_SAP_000.pdf